CLINICAL TRIAL: NCT04321031
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, DOUBLE-DUMMY, PLACEBO-CONTROLLED, DOSE-RANGING, DOSE-FINDING, PARALLEL GROUP STUDY TO ASSESS EFFICACY AND SAFETY OF PF-06865571 (DGAT2I) ALONE AND WHEN COADMINISTERED WITH PF-05221304 (ACCI) IN ADULT PARTICIPANTS WITH BIOPSY-CONFIRMED NONALCOHOLIC STEATOHEPATITIS AND FIBROSIS STAGE 2 OR 3
Brief Title: Metabolic Interventions to Resolve Non-alcoholic Steatohepatitis (NASH) With Fibrosis (MIRNA)
Acronym: MIRNA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: C2541013; 2019-004775-39 (EudraCT Number)
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis With Liver Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — ervogastat

STUDY DESIGN:
Intervention Model Description: dose ranging, dose finding
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, double dummy, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo (Placebo Comparator): participants will receive medication for 48 weeks
  Interventions: Drug: Placebo
- PF-06865571 25 milligrams (mg) twice daily (BID) (Experimental): participants will receive medication for 48 weeks
  Interventions: Drug: PF-06865571
- PF-06865571 75 mg BID (Experimental): participants will receive medication for 48 weeks
  Interventions: Drug: PF-06865571
- PF-06865571 150 mg BID (Experimental): participants will receive medication for 48 weeks
  Interventions: Drug: PF-06865571
- PF-06865571 300 mg BID (Experimental): participants will receive medication for 48 weeks
  Interventions: Drug: PF-06865571
- PF-06865571 (150 mg BID) + PF-05221304 (5 mg BID) (Experimental): participants will receive medication for 48 weeks
  Interventions: Drug: PF-06865571; Drug: PF-05221304
- PF-06865771 (300 mg BID) + PF-05221304 (10 mg BID) (Experimental): participants will receive medication for 48 weeks
  Interventions: Drug: PF-06865571; Drug: PF-05221304

INTERVENTIONS:
Drug: Placebo — Tablet
  Arms: Placebo
Drug: PF-06865571 — Tablet
  Arms: PF-06865571 (150 mg BID) + PF-05221304 (5 mg BID); PF-06865571 150 mg BID; PF-06865571 25 milligrams (mg) twice daily (BID); PF-06865571 300 mg BID; PF-06865571 75 mg BID; PF-06865771 (300 mg BID) + PF-05221304 (10 mg BID)
Drug: PF-05221304 — Tablet
  Arms: PF-06865571 (150 mg BID) + PF-05221304 (5 mg BID); PF-06865771 (300 mg BID) + PF-05221304 (10 mg BID)

SUMMARY:
The study aims to evaluate two, orally administered, investigational agents - PF-06865571 (DGAT2 inhibitor) and the coadministration of PF-06865571 with PF-05221304 (ACC inhibitor). This study is specifically designed to evaluate the effect of a range of doses of DGAT2i alone, and DGAT2i + ACCi, on resolution of NASH or improvement in liver fibrosis, as assessed histologically (via liver biopsy).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven NASH with either F2 or F3 fibrosis, per NASH CRN definition
* BMI >/= 22.5kg/m2

Exclusion Criteria:

* Evidence of other causes of liver disease such as Alcoholic steatohepatitis, (de)compensated cirrhosis, active viral hepatitis
* Any condition possibly affecting drug absorption -Unstable concomitant medical conditions, based on medical history or screening laboratory results including-
* unstable liver function tests, recent cardiovascular event(s) significant malignancies,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (290):
- United States (183):
  - Institute for Liver Health dba Arizona Liver Health, Chandler, Arizona
  - Comprehensive Interventional Care Centers (CICC), Gilbert, Arizona
  - The Institute for Liver Health, Glendale, Arizona
  - The Institute for Liver Health, Peoria, Arizona
  - Comprehensive Interventional Care Centers (CICC), Sun City, Arizona
  - Institute for Liver Health DBA Arizona Liver Health, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - Sharp Coronado Hospital, Coronado, California
  - Southern California Research Center, Coronado, California
  - Magnolia Surgery Center, El Cajon, California
  - Encino Hospital Medical Center, Encino, California
  - National Research Institute, Huntington Park, California
  - Investigational Drug Service, Altman Clinical and Translational Research Institute (ACTRI), La Jolla, California
  - University of California San Diego, Altman Clinical and Translational Research Institute Clinic, La Jolla, California
  - UCSD Altman Clinical and Transitional Research Institute, La Jolla, California
  - A V Pediatrics, Allergy & Family Medicine, Lancaster, California
  - Jatinder S. Pruthi, M.D. FACG CPI, Lancaster, California
  - Om Research LLC, Lancaster, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars-Sinai Advanced Health Sciences Pavilion (Imaging), Los Angeles, California
  - Cedars-Sinai Comprehensive Transplant Center, Los Angeles, California
  - Cedars-Sinai Medical Center Investigational Drug Services (Pharmacy), Los Angeles, California
  - S. Mark Taper Foundation Imaging Center (Liver Biopsy), Los Angeles, California
  - Providence Facey Medical Foundation, Mission Hills, California
  - Providence Holy Cross Medical Center, Mission Hills, California
  - ART Vascular, Montebello, California
  - United Medical Doctors, Murrieta, California
  - Back Bay Imaging (Liver Biopsy), Newport Beach, California
  - Advanced Imaging Center, Palmdale, California
  - Blake Wilbur Outpatient Clinic (MRI), Palo Alto, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - California Liver Research Institute, Pasadena, California
  - HMRI, Pasadena, California
  - Stanford Medicine Outpatient Center (Liver clinic/MRI), Redwood City, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Clinical Trials Research, Sacramento, California
  - Precision Research Institute, San Diego, California
  - WR-MCCR, San Diego, California
  - Sharp and Children's MRI Center, LLC, San Diego, California
  - Stanford Cancer Center South Bay (MRI), San Jose, California
  - Liberty Pacific Advanced Imaging, Tarzana, California
  - Orange County Research Center, Tustin, California
  - Upland Clinical Research, Upland, California
  - Bristol Hospital, Bristol, Connecticut
  - Bristol Radiology Center, Bristol, Connecticut
  - Connecticut Clinical Research Institute, LLC, Bristol, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Yale New Haven Hospital, Saint Raphael Campus (MRE location), New Haven, Connecticut
  - Yale Center for Clinical Investigators, Church Street South Research Unit (CSRU), New Haven, Connecticut
  - Yale Digestive Diseases (Fibroscan location), New Haven, Connecticut
  - Tower Radiology (MRI-PDFF), Brandon, Florida
  - Tower Radiology - Parsons, Brandon, Florida
  - Gastro Florida, Clearwater, Florida
  - Integrity Clinical Research, LLC, Doral, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Center for Advanced Gastroenterology, Maitland, Florida
  - Sandlake Imaging, Maitland, Florida
  - Optimus U Corporation, Miami, Florida
  - Unique Imaging (Biscayne Imaging Center), Miami, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Ivetmar Medical Group LLC, Miami, Florida
  - Vascular and Interventional Specialists of Florida (Liver Biopsy), Miami, Florida
  - Care Research Center Inc, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - TGH Imaging Powered by Tower Radiology Center (MRI), Oldsmar, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Omega Research Maitland, LLC, Orlando, Florida
  - Innovation Medical Research Center, Inc, Palmetto Bay, Florida
  - Partners Imaging Center, Sarasota, Florida
  - GCP, Global Clinical Professionals, St. Petersburg, Florida
  - Gateway (Ultrasound), St. Petersburg, Florida
  - Radiology Associates, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - AdventHealth Zephyrhills, Zephyrhills, Florida
  - Florida Medical Clinic, LLC, Zephyrhills, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Piedmont Atlanta Hospital/Piedmont Transplant Institute, Atlanta, Georgia
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Tekton Research, Inc., Snellville, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - Hendricks Regional Health, Hendricks, Indiana
  - Heartland Medical Research, Inc. (Administrative Only), Clive, Iowa
  - Iowa Digestive Disease Center, Clive, Iowa
  - Iowa Radiology, Clive, Iowa
  - MercyOne Des Moines Medical Center (Mercy Medical Center), Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Iowa Magnetic Resonance Research Facility, Iowa City, Iowa
  - Kansas Medical Clinic PA, Topeka, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Cypress Interventional, Wichita, Kansas
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Lake Charles Memorial Hospital, Lake Charles, Louisiana
  - Metropolitan Gastroenterology Associates, Marrero, Louisiana
  - Tandem Clinical Research GI, LLC, Marrero, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Gastro Health Research, Catonsville, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Michigan Clinical Research Unit (MCRU), Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - Mercy Health, Grand Rapids, Michigan
  - M1 Imaging Center, Grand Rapids, Michigan
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinical Research Center, Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Jefferson City Medical Group, P.C., Jefferson City, Missouri
  - Desert Radiology, Las Vegas, Nevada
  - Machuca Family Medicine, Las Vegas, Nevada
  - The Machuca Foundation, Inc., Las Vegas, Nevada
  - Sierra Clinical Research, Las Vegas, Nevada
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Pueblo Medical Imaging, Las Vegas, Nevada
  - Digestive Healthcare Associates, Hillsborough, New Jersey
  - University Radiology, Hillsborough, New Jersey
  - Amici Clinical Research, Raritan, New Jersey
  - Northwell Health Center for Liver Diseases, Manhasset, New York
  - Icahn School of Medicine at Mount Sinai/The Mount Sinai Hospital, New York, New York
  - M3 - Wake Research, Inc., Raleigh, North Carolina
  - Gastroenterology Associates of the Piedmont, PA, Winston-Salem, North Carolina
  - Novant Health Medical Center, Winston-Salem, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Comprehensive Diagnostic Imaging, Oklahoma City, Oklahoma
  - Digestive Disease Specialists, Inc. Endoscopy Lab, Oklahoma City, Oklahoma
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Oklahoma Spine Hospital, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC - Center for Liver Diseases at the Thomas E. Starzl Institute, Pittsburgh, Pennsylvania
  - UPMC - Center for Liver Diseases in the Digestive Disorders Clinic, Pittsburgh, Pennsylvania
  - UPMC - Translational Research Center, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Shadyside; Presbyterian Campus Pharmacy, Pittsburgh, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Roger Williams Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC- Ashley River Tower, Charleston, South Carolina
  - Chattanooga Imaging Center, Chattanooga, Tennessee
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - Vanderbilt Hepatology and Liver Transplant, Nashville, Tennessee
  - Vanderbilt University Medical Center - GI Research Office, Nashville, Tennessee
  - Vanderbilt University Medical Center - Digestive Disease Center, Nashville, Tennessee
  - Vanderbilt University Medical Center - Heart Station, Nashville, Tennessee
  - Vanderbilt University Medical Center - Interventional Radiology, Nashville, Tennessee
  - Texas Center for Interventional Surgery (Liver Biopsy Facility), Addison, Texas
  - Texas Clinical Research Institute, Arlington, Texas
  - Methodist Dallas Medical Center (MRI-PDFF), Dallas, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Touchstone Imaging, Dallas, Texas
  - Center For Diagnostic Imaging, DeSoto, Texas
  - GI Alliance, Fort Worth, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Premier Vein and Vascular, Houston, Texas
  - Centex Studies, Inc, McAllen, Texas
  - HCA Houston Healthcare Pearland, Pearland, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Diabetes and Glandular Disease Clinic, P.A., San Antonio, Texas
  - Reddy Cardiac Wellness, Sugar Land, Texas
  - Impact Research Institute, Waco, Texas
  - Gastro Health Research, Fairfax, Virginia
  - Gastro Health, LLC, Fairfax, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Sentara Leigh Hospital, Norfolk, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - VCU Medical Center Investigational Drug Service, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Gastroenterology Clinical Research, Suffolk, Virginia
  - Harborview Medical Center Investigational Drug Services, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Seattle Radiology, Seattle, Washington
  - Liver Institute Northwest, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Bulgaria (9):
  - MHAT Dr. Tota Venkova AD, Gabrovo
  - MHAT Medline Clinic AD, Plovdiv
  - Acibadem City Clinic MHAT Tokuda EAD, Sofia
  - DCC Alexandrovska EOOD, Sofia
  - UMHAT Sv. Ivan Rilski EAD, Sofia
  - UMHAT Sofiamed OOD, Sofia
  - MC New Rehabilitation Center EOOD, Stara Zagora
  - DCC Mladost-M Varna OOD, Varna
  - MC Leo Clinic EOOD, Varna
- Canada (16):
  - University of Calgary - Heritage Medical Research Clinic (HMRC), Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - Nova Scotia Health Authority QEII (Queen Elizabeth II) Health Sciences Centre, Halifax, Nova Scotia
  - Manna Research (London), London, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Resonance Magnetique du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Centre integre universitaire de sante et de services sociaux du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Ecogene-21, Chicoutimi, Quebec
  - Centre de recherche du Centre hospitalier de l'Université de Montréal (CRCHUM), Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Philips Radiation Oncology, Montreal, Quebec
  - Research Institute of the MUHC, Montreal, Quebec
  - Diex Recherche Quebec Inc., Québec
- China (14):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qingdao Central Hospital, Qingdao, Shandong
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Peking University People's Hospital, Beijing
  - Beijing YouAn Hosptial,Capital Medical University, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Tianjin Third Central Hospital, Tianjin
  - Tianjin Second People's Hospital, Tianjin
- Hong Kong (3):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
  - Alice Ho Miu Ling Nethersole Hospital, Tai Po
- India (9):
  - Surat Institute of Digestive Sciences, Surat, Gujarat
  - Gujarat Hospital - Gastro and Vascular Centre, Surat, Gujarat
  - Global Hospital - Super Speciality & Transplant Centre, Mumbai, Maharashtra
  - Max Smart Super Speciality Hospital, Saket, NEW Delhi
  - S.M.S. Medical College & Hospital, Jaipur, Rajasthan
  - Institute of Post Graduate Medical Education and Research & SSKM Hospital, Kolkata, West Bengal
  - Medanta - The Medicity, Gurugram
  - Institute of Liver and Biliary Sciences (ILBS), New Delhi
  - All India Institute of Medical Sciences (AIIMS), New Delhi
- Japan (19):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Ehime University Hospital, Tōon, Ehime
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Tokyo Medical University Ibaraki Medical Center, Inashiki-gun, Ibaraki
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Shinshu University Hospital, Matsumoto, Nagano
  - National Hospital Organization Nagasaki Medical Center, Ohmura, Nagasaki
  - Osaka Rosai Hospital, Sakai, Osaka
  - Saiseikai Suita Hospital, Suita, Osaka
  - Juntendo University Shizuoka Hospital, Izunokuni, Shizuoka
  - Chiba University Hospital, Chiba
  - Fukui-Ken Saiseikai Hospital, Fukui
  - Gifu Municipal Hospital, Gifu
  - Kagoshima University Hospital, Kagoshima
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Miyazaki Medical Center Hospital, Miyazaki
  - Saga University Hospital, Saga
  - Yamagata University Hospital, Yamagata
- Poland (13):
  - Szpital Zakonu Bonifratrow, Katowice
  - NZOZ Vita Longa Sp. z o.o., Katowice
  - Uniwersyteckie Centrum Kliniczne im. prof. K. Gibinskiego Slaskiego Uniwersytetu Medycznego, Katowice
  - Orthos Szpital Wielospecjalistyczny Sp. z o.o. (Liver Biopsy), Komorowice
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Szpital Zakonu Bonifratrów św. Jana Grandego w Krakowie sp. z o.o. (Liver Biopsy), Krakow
  - Krakowskie Centrum Medyczne, Krakow
  - Wojewodzki Specjalistyczny Szpital im. Dr. Wl. Bieganskiego w Lodzi, Lodz
  - ID Clinic, Mysłowice
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Futuremeds Sp. z o.o., Wroclaw
  - ETG Zamosc, Zamość
  - Samodzielny Publiczny Szpital Wojewodzki im. Papieza Jana Pawla II, Zamość
- Puerto Rico (4):
  - Clinical Research Puerto Rico, San Juan
  - Latin Clinical Trial Center, San Juan
  - GCM Medical Group PSC, San Juan
  - FDI Clinical Research, San Juan
- Slovakia (8):
  - Fakultna nemocnica s poliklinikou F. D. Roosevelta Banska Bystrica, Banská Bystrica
  - Medispektrum, s.r.o, Bratislava
  - SUMMIT CLINICAL RESEARCH, s.r.o., Bratislava - Mestska Cast Nove Mesto
  - Lama Medical Care s.r.o., Bratislava - Mestska Cast Ruzinov
  - Univerzitna nemocnica L. Pasteura Kosice, Kosice - Mestska Cast Zapad
  - KM Management spol. s.r.o., Gastroenterologicke a hepatologicke centrum Nitra, Nitra
  - Fakultna nemocnica Nitra, Nitra
  - JAL, s.r.o., Trnava
- South Korea (5):
  - SMG-SNU Boramae Medical Center, Dongjak-gu, Seoul
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Severance Hospital Yonsei University Health System, Seoul
- Taiwan (7):
  - Changhua Christian Hospital, Changhua, Changhua County
  - Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University (NCKU) Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Wong VW, Amin NB, Takahashi H, Darekar A, Tacke F, Kiszko J, Rodriguez H, Nakajima A, Alkhouri N, Charlton M, Anstee QM. Efficacy and safety of ervogastat alone and in combination with clesacostat in patients with biopsy-confirmed metabolic dysfunction-associated steatohepatitis and F2-F3 fibrosis (MIRNA): results from a phase 2, randomised, double-blind, double-dummy study. Lancet Gastroenterol Hepatol. 2025 Oct;10(10):924-940. doi: 10.1016/S2468-1253(25)00128-1. Epub 2025 Jul 31. PMID 40753985
- [Derived] Amin NB, Darekar A, Anstee QM, Wong VW, Tacke F, Vourvahis M, Lee DS, Charlton M, Alkhouri N, Nakajima A, Yunis C. Efficacy and safety of an orally administered DGAT2 inhibitor alone or coadministered with a liver-targeted ACC inhibitor in adults with non-alcoholic steatohepatitis (NASH): rationale and design of the phase II, dose-ranging, dose-finding, randomised, placebo-controlled MIRNA (Metabolic Interventions to Resolve NASH with fibrosis) study. BMJ Open. 2022 Mar 30;12(3):e056159. doi: 10.1136/bmjopen-2021-056159. PMID 35354614
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2541013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 256 participants with biopsy confirmed Non-alcoholic Steatohepatitis (NASH) with fibrosis state (F2-F3) were randomized, of which 255 were treated.
Pre-assignment Details: F2: significant stage of fibrosis when scarring had occurred and extended outside liver area and F3: severe stage of fibrosis with spreading and forming bridges with other fibrotic liver areas.
Groups:
- Placebo: Participants were randomized to receive 2 tablets of diacylglycerol acyltransferase 2 inhibitor (PF-06865571/DGAT2i) matching placebo and 1 tablet of acetyl-CoA carboxylase inhibitor (PF-05221304/ACCi) matching placebo twice a day (BID) for 48 weeks by oral administration. Participants were followed up to 52 weeks.
- DGAT2i/PF-06865571 25 mg BID: Participants were randomized to receive 1 tablet of DGAT2i 25 milligrams (mg) along with 1 tablet of DGAT2i and ACCi matching placebo BID for 48 weeks by oral administration. Participants were followed up to 52 weeks.
- DGAT2i/PF-06865571 75 mg BID: Participants were randomized to receive 1 tablet of DGAT2i 25 mg, 1 tablet of DGAT2i 50 mg and 1 tablet of ACCi matching placebo BID for 48 weeks by oral administration. Participants were followed up to 52 weeks.
- DGAT2i/PF-06865571 150 mg BID: Participants were randomized to receive 1 tablet of DGAT2i matching placebo, 1 tablet of DGAT2i 150 mg and 1 tablet of ACCi matching placebo BID for 48 weeks by oral administration. Participants were followed up to 52 weeks.
- DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID: Participants were randomized to receive 1 tablet of DGAT2i matching placebo, 1 tablet of DGAT2i 150 mg and 1 tablet of ACCi 5 mg BID for 48 weeks by oral administration. Participants were followed up to 52 weeks.
- DGAT2i/PF-06865571 300 mg BID: Participants were randomized to receive 2 tablets of DGAT2i 150 mg and 1 tablet of ACCi matching placebo BID for 48 weeks by oral administration. Participants were followed up to 52 weeks.
- DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID: Participants were randomized to receive 2 tablets of DGAT2i 150 mg and 1 tablet of ACCi 10 mg BID for 48 weeks by oral administration. Participants were followed up to 52 weeks.
Period: Overall Study
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID
Started | 34 | 35 | 48 | 42 | 35 | 31 | 30
Completed | 32 | 31 | 45 | 35 | 32 | 26 | 28
Not Completed | 2 | 4 | 3 | 7 | 3 | 5 | 2
Not completed — Adverse Event | 0 | 2 | 2 | 2 | 2 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 3 | 1 | 0 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who took at least 1 dose of investigational product. Participants were analyzed according to the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID | Total
Number analyzed (Participants) | 34 | 35 | 48 | 42 | 35 | 31 | 30 | 255
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.21 (12.00) | 56.54 (11.38) | 56.02 (12.67) | 55.95 (11.32) | 56.60 (10.23) | 59.65 (7.49) | 54.23 (11.32) | 56.28 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 31 | 28 | 24 | 20 | 15 | 154
  Male | 17 | 16 | 17 | 14 | 11 | 11 | 15 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 8 | 15 | 13 | 10 | 6 | 11 | 8 | 71
  Ethnicity: Not Hispanic or Latino | 24 | 20 | 35 | 29 | 29 | 18 | 20 | 175
  Ethnicity: Unknown or Not Reported | 2 | 0 | 0 | 3 | 0 | 2 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Race: Asian | 12 | 10 | 16 | 14 | 13 | 11 | 11 | 87
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Race: Black or African American | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 5
  Race: White | 21 | 20 | 31 | 24 | 19 | 17 | 18 | 150
  Race: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Race: Unknown or Not Reported | 1 | 3 | 1 | 3 | 2 | 2 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Proportion of Participants Achieving Resolution of NASH Without Worsening/Improvement of Fibrosis by >=1 Stage Without Worsening of NASH/Both Based on Assessment by Sponsor-Identified Central Pathologist at Week 48:Bayesian Dose Response Model (BDRM)
Description: NASH resolution: disappearance of ballooning (Nonalcoholic Fatty Liver Disease [NAFLD] Activity Score [NAS] ballooning score=0;0=no ballooning,1=few balloon cells,2=many cells with prominent ballooning; higher scores(HS)=more disease activity [DA]),residual/no lobular inflammation(NAS lobular inflammation score 0/1,0=no foci,1= <2 foci, 2=2-4 foci,3= >4 foci; HS=more DA),NAS steatosis score 0,1,2,3; 0= <5% hepatocytes involved (HI),1=5-33% HI ,2= 34-66% HI, 3= >66% HI; HS=more DA. No worsening of fibrosis: no change/decrease of at least 1 stage in Brunt-Kleiner scale (BKS) compared to baseline (CTB). Improvement in fibrosis by >=1 stage: decrease of at least 1 stage in BKS CTB. No worsening of NASH: no change/increase in NAS for ballooning, inflammation, steatosis CTB. BDRM utilized to characterize dose response across BID treatment groups, estimate posterior mean proportion (& 90% credible interval [CI], indicated as 'confidence interval' below) for placebo and each BID dose studied.
Time Frame: Week 48
Population: BKS: scaling for fibrosis (0=none,1=perisinusoidal/ periportal,2=perisinusoidal, portal/ periportal,3=bridging,4=cirrhosis; higher scores=more DA). Full analysis set (FAS):all randomized participants who took at least 1 dose of investigational product who had provided baseline data for primary endpoint. This outcome measure was not planned to be analyzed in combination arms (DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID and DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID).
Measure: Mean (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 300 mg BID
Number analyzed (Participants) | 34 | 35 | 48 | 42 | 31
Proportion of participants | 0.38 [0.26 to 0.50] | 0.45 [0.38 to 0.53] | 0.48 [0.42 to 0.55] | 0.50 [0.43 to 0.57] | 0.51 [0.43 to 0.59]
Statistical Analysis 1: Comparison: Placebo vs DGAT2i/PF-06865571 25 mg BID; The model was applied to the raw number of responders and non-responders utilizing a Bayesian methodology approach with non-informative priors as described in the statistical analysis plan (SAP); Test type: Superiority; Risk Difference (RD) = 0.08, 90% CI 2-sided [-0.02 to 0.20] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 2: Comparison: Placebo vs DGAT2i/PF-06865571 75 mg BID; The model was applied to the raw number of responders and non-responders utilizing a Bayesian methodology approach with non-informative priors as described in the SAP; Test type: Superiority; Risk Difference (RD) = 0.10, 90% CI 2-sided [-0.03 to 0.24] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 3: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.12, 90% CI 2-sided [-0.03 to 0.26] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 4: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.13, 90% CI 2-sided [-0.04 to 0.28] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval

2. Primary Outcome: Number of Participants Achieving Resolution of NASH Without Worsening or Improvement in Fibrosis by >= 1 Stage Without Worsening of NASH or Both Based on Assessment by Sponsor-Identified Central Pathologist at Week 48: Logistic Regression Model
Description: Resolution of NASH: disappearance of ballooning (NAS ballooning score= 0; where 0= no ballooning, 1= few balloon cells, 2= many cells with prominent ballooning; higher scores= more disease activity), residual or no lobular inflammation (NAS lobular inflammation score 0 or 1, where 0= no foci, 1= <2 foci, 2= 2-4 foci, 3= >4 foci; higher scores= more disease activity), NAS steatosis score 0, 1, 2, or 3, where 0= <5% hepatocytes involved, 1= 5-33% hepatocytes involved, 2= 34-66% hepatocytes involved, 3= >66% hepatocytes involved; higher scores= more disease activity. No worsening of fibrosis: no change or decrease of at least 1 stage in BKS compared to baseline. Improvement in fibrosis by >=1 stage: decrease of at least 1 stage in BKS compared to baseline. No worsening of NASH: no change or increase in NAS for ballooning, inflammation, steatosis compared to baseline.
Time Frame: Week 48
Population: BKS: scaling for fibrosis (0= none, 1= perisinusoidal/ periportal, 2= perisinusoidal, portal/periportal, 3= bridging, 4= cirrhosis; higher scores= more disease activity). Logistic Regression model included treatment and baseline F2/F3 as factors. Full analysis set included all randomized participants who took at least 1 dose of investigational product who had provided baseline data for the primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID
Number analyzed (Participants) | 34 | 35 | 48 | 42 | 35 | 31 | 30
Participants | 13 [NA to NA] | 16 [0.61 to 3.05] | 25 [0.83 to 3.72] | 21 [0.74 to 3.48] | 23 [1.35 to 7.04] | 14 [0.58 to 3.08] | 19 [1.19 to 6.56]
Statistical Analysis 1: Comparison: Placebo vs DGAT2i/PF-06865571 75 mg BID; Risk difference and 2-sided 90% confidence interval for risk difference were calculated by using the observed placebo/corresponding BID rate and estimated odds ratio from the logistic regression model; Test type: Superiority; Risk Difference (RD) = 0.14, 90% CI 2-sided [-0.04 to 0.32]
Statistical Analysis 2: Comparison: Placebo vs DGAT2i/PF-06865571 25 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.08, 90% CI 2-sided [-0.11 to 0.27]
Statistical Analysis 3: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.12, 90% CI 2-sided [-0.07 to 0.30]
Statistical Analysis 4: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.27, 90% CI 2-sided [0.07 to 0.43]
Statistical Analysis 5: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.07, 90% CI 2-sided [-0.12 to 0.27]
Statistical Analysis 6: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.25, 90% CI 2-sided [0.04 to 0.42]
Statistical Analysis 7: Comparison: DGAT2i/PF-06865571 150 mg BID vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; Risk difference and 2-sided 50% confidence interval for risk difference were calculated by using the observed placebo/corresponding BID rate and estimated odds ratio from the logistic regression model; Test type: Superiority; Risk Difference (RD) = 0.16, 50% CI 2-sided [0.08 to 0.23]
Statistical Analysis 8: Comparison: DGAT2i/PF-06865571 150 mg BID vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.16, 90% CI 2-sided [-0.03 to 0.31]
Statistical Analysis 9: Comparison: DGAT2i/PF-06865571 300 mg BID vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Risk Difference (RD) = 0.18, 50% CI 2-sided [0.09 to 0.26]
Statistical Analysis 10: Comparison: DGAT2i/PF-06865571 300 mg BID vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.18, 90% CI 2-sided [-0.03 to 0.35]

3. Secondary Outcome: Percent Change From Baseline in Liver Fat at Week 48: Bayesian Dose Response Model
Description: Magnetic resonance imaging proton density fat fraction (MRI-PDFF) is an established method that enables quantification of fat content in the liver.
Time Frame: Baseline, Week 48
Population: Full analysis set: all randomized participants who took at least 1 dose of investigational product who had provided baseline data for primary endpoint. This outcome measure was not planned to be analyzed in combination arms (DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID and DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID). Here, ''Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Mean (90% Confidence Interval); unit: Percent change
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 300 mg BID
Number analyzed (Participants) | 15 | 14 | 21 | 18 | 11
Percent change | -10.79 [-38.30 to 18.99] | -36.76 [-52.57 to -20.15] | -46.20 [-59.64 to -32.82] | -51.33 [-66.78 to -36.59] | -55.53 [-77.23 to -37.64]
Statistical Analysis 1: Comparison: Placebo vs DGAT2i/PF-06865571 25 mg BID; Test type: Superiority; Least Square (LS) Mean = -25.98, 90% CI 2-sided [-58.42 to -2.57]
Statistical Analysis 2: Comparison: Placebo vs DGAT2i/PF-06865571 75 mg BID; Test type: Superiority; LS Mean = -35.41, 90% CI 2-sided [-69.41 to -5.42]
Statistical Analysis 3: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID; Test type: Superiority; LS Mean = -40.54, 90% CI 2-sided [-75.55 to -7.32]
Statistical Analysis 4: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID; Test type: Superiority; LS Mean = -44.74, 90% CI 2-sided [-81.72 to -8.42]

4. Secondary Outcome: Percent Change From Baseline in Liver Fat at Week 48: Pairwise Comparisons With Analysis of Covariance (ANCOVA)
Description: MRI-PDFF is an established method that enables quantification of fat content in the liver.
Time Frame: Baseline, Week 48
Population: Full analysis set: all randomized participants who took at least 1 dose of investigational product who had provided baseline data for primary endpoint. Here, ''Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID
Number analyzed (Participants) | 9 | 12 | 18 | 12 | 11 | 8 | 8
Percent change | 1.41 (22.11) | -41.00 (18.89) | -42.53 (15.66) | -58.77 (19.44) | -67.76 (19.93) | -49.76 (23.70) | -68.83 (23.72)
Statistical Analysis 1: Comparison: Placebo vs DGAT2i/PF-06865571 25 mg BID; Log-transformed relative changes from baseline are modelled using an ANCOVA model with treatment and baseline fibrosis stage (F2/F3) as factors, and log-transformed baseline liver fat as a covariate; Test type: Superiority; LS Mean = -41.82, 90% CI 2-sided [-62.57 to -9.57]
Statistical Analysis 2: Comparison: Placebo vs DGAT2i/PF-06865571 75 mg BID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; LS Mean = -43.33, 90% CI 2-sided [-62.37 to -14.64]
Statistical Analysis 3: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; LS Mean = -59.35, 90% CI 2-sided [-73.95 to -36.55]
Statistical Analysis 4: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; LS Mean = -68.21, 90% CI 2-sided [-79.72 to -50.15]
Statistical Analysis 5: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; LS Mean = -50.46, 90% CI 2-sided [-69.53 to -19.44]
Statistical Analysis 6: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; LS Mean = -69.27, 90% CI 2-sided [-81.08 to -50.07]
Statistical Analysis 7: Comparison: DGAT2i/PF-06865571 150 mg BID vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; LS Mean = -21.80, 50% CI 2-sided [-34.02 to -7.32]
Statistical Analysis 8: Comparison: DGAT2i/PF-06865571 150 mg BID vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; LS Mean = -21.80, 90% CI 2-sided [-48.51 to 18.76]
Statistical Analysis 9: Comparison: DGAT2i/PF-06865571 300 mg BID vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; LS Mean = -37.97, 50% CI 2-sided [-49.40 to -23.95]
Statistical Analysis 10: Comparison: DGAT2i/PF-06865571 300 mg BID vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; LS Mean = -37.97, 90% CI 2-sided [-62.41 to 2.37]

5. Secondary Outcome: Mean Proportion of Participants Achieving Resolution of NASH, Without Worsening of Fibrosis Based on Assessment by Sponsor-Identified Central Pathologist(s) at Week 48: Bayesian Dose Response Model
Description: Resolution of NASH: disappearance of ballooning (NAS ballooning score= 0; where 0= no ballooning, 1= few balloon cells, 2= many cells with prominent ballooning; higher scores= more disease activity), residual or no lobular inflammation (NAS lobular inflammation score 0 or 1, where 0= no foci, 1= <2 foci, 2= 2-4 foci, 3= >4 foci; higher scores= more disease activity), NAS steatosis score 0, 1, 2 or 3, where 0= <5% HI, 1= 5-33% HI, 2= 34-66% HI, 3= >66% HI; higher scores= more disease activity. No worsening of fibrosis: no change or decrease of at least 1 stage in BKS compared to baseline. BKS: scaling for fibrosis (0= none, 1= perisinusoidal/ periportal, 2= perisinusoidal, portal/ periportal, 3= bridging, 4= cirrhosis; higher scores= more disease activity). BDRM utilized to characterize dose response across BID treatment groups, estimate posterior mean proportion (& 90% credible interval [CI], indicated as 'confidence interval' below) for placebo and each BID dose studied.
Time Frame: Week 48
Population: FAS included all randomized participants who took at least 1 dose of investigational product who had provided baseline data for primary endpoint. This outcome measure was not planned to be analyzed in combination arms (DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID and DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID).
Measure: Mean (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 300 mg BID
Number analyzed (Participants) | 34 | 35 | 48 | 42 | 31
Proportion of participants | 0.11 [0.04 to 0.20] | 0.32 [0.23 to 0.40] | 0.37 [0.31 to 0.44] | 0.40 [0.33 to 0.47] | 0.41 [0.34 to 0.50]
Statistical Analysis 1: Comparison: Placebo vs DGAT2i/PF-06865571 25 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.21, 90% CI 2-sided [0.09 to 0.32] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 2: Comparison: Placebo vs DGAT2i/PF-06865571 75 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.27, 90% CI 2-sided [0.15 to 0.37] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 3: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.29, 90% CI 2-sided [0.18 to 0.39] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 4: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.31, 90% CI 2-sided [0.19 to 0.42] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval

6. Secondary Outcome: Number of Participants Achieving Resolution of NASH, Without Worsening of Fibrosis Based on Assessment by Sponsor-Identified Central Pathologist(s) at Week 48: Pairwise Comparisons With Logistic Regression Model
Description: Resolution of NASH: disappearance of ballooning (NAS ballooning score= 0; where 0= no ballooning, 1= few balloon cells, 2= many cells with prominent ballooning; higher scores= more disease activity), residual or no lobular inflammation (NAS lobular inflammation score 0 or 1, where 0= no foci, 1= <2 foci, 2= 2-4 foci, 3= >4 foci; higher scores= more disease activity), NAS steatosis score 0, 1, 2 or 3, where 0= <5% hepatocytes involved, 1= 5-33% hepatocytes involved, 2= 34-66% hepatocytes involved, 3= >66% hepatocytes involved; higher scores= more disease activity. No worsening of fibrosis: no change or decrease of at least 1 stage in Brunt-Kleiner scale compared to baseline. Brunt-Kleiner scale included scaling for fibrosis (0= none, 1= perisinusoidal/ periportal, 2= perisinusoidal, portal/ periportal, 3= bridging, 4= cirrhosis; higher scores = more disease activity). Logistic Regression model included treatment and baseline fibrosis stage (F2/F3) as factors.
Time Frame: Week 48
Population: Full analysis set included all randomized participants who took at least 1 dose of investigational product who had provided baseline data for primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID
Number analyzed (Participants) | 34 | 35 | 48 | 42 | 35 | 31 | 30
Participants | 3 | 11 | 22 | 13 | 22 | 13 | 17
Statistical Analysis 1: Comparison: Placebo vs DGAT2i/PF-06865571 25 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.23, 90% CI 2-sided [0.04 to 0.51]
Statistical Analysis 2: Comparison: Placebo vs DGAT2i/PF-06865571 75 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.37, 90% CI 2-sided [0.13 to 0.63]
Statistical Analysis 3: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.22, 90% CI 2-sided [0.04 to 0.49]
Statistical Analysis 4: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.54, 90% CI 2-sided [0.26 to 0.75]
Statistical Analysis 5: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.34, 90% CI 2-sided [0.10 to 0.61]
Statistical Analysis 6: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.48, 90% CI 2-sided [0.20 to 0.72]
Statistical Analysis 7: Comparison: DGAT2i/PF-06865571 150 mg BID vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Risk Difference (RD) = 0.32, 50% CI 2-sided [0.24 to 0.39]
Statistical Analysis 8: Comparison: DGAT2i/PF-06865571 150 mg BID vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.32, 90% CI 2-sided [0.12 to 0.48]
Statistical Analysis 9: Comparison: DGAT2i/PF-06865571 300 mg BID vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Risk Difference (RD) = 0.14, 50% CI 2-sided [0.06 to 0.23]
Statistical Analysis 10: Comparison: DGAT2i/PF-06865571 300 mg BID vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.14, 90% CI 2-sided [-0.06 to 0.33]

7. Secondary Outcome: Mean Proportion of Participants Achieving Improvement in Fibrosis by >=1 Stage, Without Worsening of NASH Based on Assessment by Sponsor-Identified Central Pathologist(s) at Week 48: Bayesian Dose Response Model
Description: Improvement in fibrosis by >=1 stage: decrease of at least 1 stage in Brunt-Kleiner scale compared to baseline. No worsening of fibrosis: no change or decrease of at least 1 stage in Brunt-Kleiner scale compared to baseline. Brunt-Kleiner scale included scaling for fibrosis (0= none, 1= perisinusoidal/ periportal, 2= perisinusoidal, portal/ periportal, 3= bridging, 4= cirrhosis; higher scores = more disease activity). BDRM utilized to characterize dose response across BID treatment groups, estimate posterior mean proportion (& 90% credible interval [CI], indicated as 'confidence interval' below) for placebo and each BID dose studied.
Time Frame: Week 48
Population: Full analysis set included all randomized participants who took at least 1 dose of investigational product who had provided baseline data for primary endpoint. This outcome measure was not planned to be analyzed in combination arms (DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID and DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID).
Measure: Mean (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 300 mg BID
Number analyzed (Participants) | 34 | 35 | 48 | 42 | 31
Proportion of participants | 0.33 [0.22 to 0.45] | 0.28 [0.21 to 0.35] | 0.25 [0.20 to 0.31] | 0.24 [0.18 to 0.30] | 0.22 [0.14 to 0.30]
Statistical Analysis 1: Comparison: Placebo vs DGAT2i/PF-06865571 25 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = -0.05, 90% CI 2-sided [-0.16 to 0.02] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 2: Comparison: Placebo vs DGAT2i/PF-06865571 75 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = -0.07, 90% CI 2-sided [-0.20 to 0.03] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 3: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = -0.09, 90% CI 2-sided [-0.23 to 0.04] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 4: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = -0.10, 90% CI 2-sided [-0.26 to 0.05] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval

8. Secondary Outcome: Number of Participants Achieving Improvement in Fibrosis by >=1 Stage, Without Worsening of NASH Based on Assessment by Sponsor-Identified Central Pathologist(s) at Week 48: Pairwise Comparisons With Logistic Regression Model
Description: Improvement in fibrosis by >=1 stage: decrease of at least 1 stage in Brunt-Kleiner scale compared to baseline. No worsening of fibrosis: no change/decrease of at least 1 stage in Brunt-Kleiner scale compared to baseline. Brunt-Kleiner scale included scaling for fibrosis (0= none, 1= perisinusoidal/ periportal, 2= perisinusoidal, portal/ periportal, 3= bridging, 4= cirrhosis; higher scores = more DA). Logistic Regression model included treatment and baseline fibrosis stage (F2/F3) as factors.
Time Frame: Week 48
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID: Participants were randomized to receive 1 tablet of DGAT2i matching placebo, 1 tablet of DGAT2i 150 mg and 1 tablet of ACCi 5 mg BID for 48 weeks by oral administration. Participants were followed up up to 52 weeks.
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID
Number analyzed (Participants) | 34 | 35 | 48 | 42 | 35 | 31 | 30
Participants | 12 | 10 | 10 | 14 | 13 | 4 | 12
Statistical Analysis 1: Comparison: Placebo vs DGAT2i/PF-06865571 25 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = -0.07, 90% CI 2-sided [-0.21 to 0.13]
Statistical Analysis 2: Comparison: Placebo vs DGAT2i/PF-06865571 75 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = -0.14, 90% CI 2-sided [-0.25 to 0.02]
Statistical Analysis 3: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = -0.02, 90% CI 2-sided [-0.17 to 0.17]
Statistical Analysis 4: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.02, 90% CI 2-sided [-0.15 to 0.22]
Statistical Analysis 5: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = -0.22, 90% CI 2-sided [-0.30 to -0.05]
Statistical Analysis 6: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.05, 90% CI 2-sided [-0.13 to 0.26]
Statistical Analysis 7: Comparison: DGAT2i/PF-06865571 150 mg BID vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Risk Difference (RD) = 0.04, 50% CI 2-sided [-0.03 to 0.12]
Statistical Analysis 8: Comparison: DGAT2i/PF-06865571 150 mg BID vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.04, 90% CI 2-sided [-0.12 to 0.23]
Statistical Analysis 9: Comparison: DGAT2i/PF-06865571 300 mg BID vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Risk Difference (RD) = 0.27, 50% CI 2-sided [0.17 to 0.38]
Statistical Analysis 10: Comparison: DGAT2i/PF-06865571 300 mg BID vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.27, 90% CI 2-sided [0.06 to 0.53]

9. Secondary Outcome: Mean Proportion of Participants Achieving Improvement in Fibrosis by >=2 Stage, Without Worsening of NASH Based on Assessment by Sponsor-Identified Central Pathologist(s) at Week 48: Bayesian Dose Response Model
Description: Improvement in fibrosis by >=2 stage: decrease of at least 2 points in total NAS compared to baseline, without progression of fibrosis. No worsening of NASH: no change or no increase in NAS for ballooning (NAS ballooning score= 0; where 0= no ballooning, 1= few balloon cells, 2= many cells with prominent ballooning; higher scores= more disease activity), inflammation (NAS lobular inflammation score 0 or 1, where 0= no foci, 1= <2 foci, 2= 2-4 foci, 3= >4 foci; higher scores= more disease activity), steatosis (NAS steatosis score 0, 1, 2, or 3, where 0= <5% hepatocytes involved, 1= 5-33% hepatocytes involved, 2= 34-66% hepatocytes involved, 3= >66% hepatocytes involved; higher scores=more disease activity) compared to baseline. BDRM utilized to characterize dose response across BID treatment groups, estimate posterior mean proportion (& 90% credible interval [CI], indicated as 'confidence interval' below) for placebo and each BID dose studied.
Time Frame: Week 48
Population: as for outcome 7
Measure: Mean (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 300 mg BID
Number analyzed (Participants) | 34 | 35 | 48 | 42 | 31
Proportion of participants | 0.05 [0.01 to 0.10] | 0.08 [0.04 to 0.11] | 0.09 [0.05 to 0.12] | 0.09 [0.06 to 0.14] | 0.10 [0.06 to 0.16]
Statistical Analysis 1: Comparison: Placebo vs DGAT2i/PF-06865571 25 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.03, 90% CI 2-sided [-0.01 to 0.08] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 2: Comparison: Placebo vs DGAT2i/PF-06865571 75 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.04, 90% CI 2-sided [-0.02 to 0.09] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 3: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.05, 90% CI 2-sided [-0.02 to 0.11] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 4: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.05, 90% CI 2-sided [-0.02 to 0.12] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval

10. Secondary Outcome: Number of Participants Achieving Improvement in Fibrosis by >=2 Stage, Without Worsening of NASH Based on Assessment by Sponsor-Identified Central Pathologist(s) at Week 48: Pairwise Comparisons With Logistic Regression Model
Description: Improvement in fibrosis by >=2 stage: decrease of at least 2 points in total NAS compared to baseline, without progression of fibrosis. No worsening of NASH: no change or no increase in NAS for ballooning (NAS ballooning score= 0; where 0= no ballooning, 1= few balloon cells, 2= many cells with prominent ballooning; higher scores= more disease activity), inflammation (NAS lobular inflammation score 0 or 1, where 0= no foci, 1= <2 foci, 2= 2-4 foci, 3= >4 foci; higher scores= more disease activity), steatosis (NAS steatosis score 0, 1, 2 or 3, where 0= <5% hepatocytes involved, 1= 5-33% hepatocytes involved, 2= 34-66% hepatocytes involved, 3= >66% hepatocytes involved; higher scores= more disease activity) compared to baseline. Logistic Regression model included treatment and baseline fibrosis stage (F2/F3) as factors.
Time Frame: Week 48
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID
Number analyzed (Participants) | 34 | 35 | 48 | 42 | 35 | 31 | 30
Participants | 1 | 4 | 3 | 5 | 7 | 2 | 6
Statistical Analysis 1: Comparison: Placebo vs DGAT2i/PF-06865571 25 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.09, 90% CI 2-sided [-0.01 to 0.43]
Statistical Analysis 2: Comparison: Placebo vs DGAT2i/PF-06865571 75 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.03, 90% CI 2-sided [-0.02 to 0.29]
Statistical Analysis 3: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.09, 90% CI 2-sided [-0.01 to 0.43]
Statistical Analysis 4: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.17, 90% CI 2-sided [0.01 to 0.57]
Statistical Analysis 5: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.04, 90% CI 2-sided [-0.02 to 0.33]
Statistical Analysis 6: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.17, 90% CI 2-sided [0.01 to 0.58]
Statistical Analysis 7: Comparison: DGAT2i/PF-06865571 150 mg BID vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Risk Difference (RD) = 0.08, 50% CI 2-sided [0.02 to 0.16]
Statistical Analysis 8: Comparison: DGAT2i/PF-06865571 150 mg BID vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.08, 90% CI 2-sided [-0.04 to 0.30]
Statistical Analysis 9: Comparison: DGAT2i/PF-06865571 300 mg BID vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Risk Difference (RD) = 0.13, 50% CI 2-sided [0.06 to 0.24]
Statistical Analysis 10: Comparison: DGAT2i/PF-06865571 300 mg BID vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.13, 90% CI 2-sided [-0.01 to 0.44]

11. Secondary Outcome: Mean Proportion of Participants Achieving Improvement of >=2 Points in Total NAS, Without Progression of Fibrosis Based on Assessment by Sponsor-Identified Central Pathologist(s) at Week 48: Bayesian Dose Response Model
Description: Improvement of >=2 points in Total NAS: decrease of at least 2 points in Total NAS compared to baseline, without progression of fibrosis. Total NAS ranged 0 to 8, higher scores= more disease activity and calculated as sum of scores of steatosis (0= <5% hepatocytes involved, 1=5-33% hepatocytes involved, 2=34-66% hepatocytes involved, 3= >66% hepatocytes involved; higher scores= more disease activity), lobular inflammation (0= no foci, 1= <2 foci, 2= 2-4 foci, 3= >4 foci; higher scores= more disease activity), ballooning (0= no ballooning, 1= few balloon cells, 2= many cells with prominent ballooning; higher scores= more disease activity). If sub-scale scores non evaluable or missing, total score was derived as missing. BDRM utilized to characterize dose response across BID treatment groups, estimate posterior mean proportion (& 90% credible interval [CI], indicated as 'confidence interval' below) for placebo and each BID dose studied.
Time Frame: Week 48
Population: as for outcome 7
Measure: Mean (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 300 mg BID
Number analyzed (Participants) | 34 | 35 | 48 | 42 | 31
Proportion of participants | 0.24 [0.13 to 0.37] | 0.42 [0.33 to 0.50] | 0.47 [0.40 to 0.54] | 0.49 [0.42 to 0.57] | 0.51 [0.43 to 0.59]
Statistical Analysis 1: Comparison: Placebo vs DGAT2i/PF-06865571 25 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.18, 90% CI 2-sided [0.05 to 0.31] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 2: Comparison: Placebo vs DGAT2i/PF-06865571 75 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.23, 90% CI 2-sided [0.09 to 0.36] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 3: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.25, 90% CI 2-sided [0.10 to 0.38] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval
Statistical Analysis 4: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Difference (RD) = 0.27, 90% CI 2-sided [0.11 to 0.40] — Reported values reflect a 90% Credible Interval rather than a 90% Confidence Interval

12. Secondary Outcome: Number of Participants Achieving Improvement of >=2 Points in Total NAS Without Progression of Fibrosis Based on Assessment by Sponsor-Identified Central Pathologist(s) at Week 48: Pairwise Comparisons With Logistic Regression Model
Description: Improvement of >=2 points in Total NAS: decrease of at least 2 points in Total NAS compared to baseline, without progression of fibrosis. Total NAS ranged from 0 to 8, higher scores= more DA and calculated as sum of scores of steatosis (0= <5% hepatocytes involved, 1= 5-33% hepatocytes involved, 2= 34-66% hepatocytes involved, 3= >66% hepatocytes involved; higher scores= more DA), lobular inflammation (0= no foci, 1= <2 foci, 2= 2-4 foci, 3= >4 foci; higher scores= more DA), ballooning (0= no ballooning, 1= few balloon cells, 2= many cells with prominent ballooning; higher scores= more DA). If any of the sub-scale scores were non evaluable/missing, then the total score was derived as missing. Logistic Regression model included treatment and baseline fibrosis stage (F2/F3) as factors.
Time Frame: Week 48
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID
Number analyzed (Participants) | 34 | 35 | 48 | 42 | 35 | 31 | 30
Participants | 8 | 13 | 28 | 21 | 25 | 12 | 19
Statistical Analysis 1: Comparison: Placebo vs DGAT2i/PF-06865571 25 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.14, 90% CI 2-sided [-0.04 to 0.36]
Statistical Analysis 2: Comparison: Placebo vs DGAT2i/PF-06865571 75 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.35, 90% CI 2-sided [0.15 to 0.53]
Statistical Analysis 3: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.26, 90% CI 2-sided [0.06 to 0.46]
Statistical Analysis 4: Comparison: Placebo vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.48, 90% CI 2-sided [0.27 to 0.63]
Statistical Analysis 5: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.16, 90% CI 2-sided [-0.03 to 0.38]
Statistical Analysis 6: Comparison: Placebo vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.40, 90% CI 2-sided [0.18 to 0.58]
Statistical Analysis 7: Comparison: DGAT2i/PF-06865571 150 mg BID vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Risk Difference (RD) = 0.22, 50% CI 2-sided [0.15 to 0.28]
Statistical Analysis 8: Comparison: DGAT2i/PF-06865571 150 mg BID vs DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.22, 90% CI 2-sided [0.03 to 0.35]
Statistical Analysis 9: Comparison: DGAT2i/PF-06865571 300 mg BID vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; Risk Difference (RD) = 0.24, 50% CI 2-sided [0.16 to 0.32]
Statistical Analysis 10: Comparison: DGAT2i/PF-06865571 300 mg BID vs DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Risk Difference (RD) = 0.24, 90% CI 2-sided [0.03 to 0.42]

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant/ clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Serious adverse events (SAE) was any untoward medical occurrence at any dose that: resulted in death, was life threatening (risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect. AEs included both serious and all non-serious AEs. TEAEs were defined as newly occurring or worsening AE after the first dose of study drug.
Time Frame: From first dose of study drug (Day 1) up to 4 weeks after last dose of study drug (maximum up to approximately 52 weeks)
Population: Safety population included all participants who took at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID
Number analyzed (Participants) | 34 | 35 | 48 | 42 | 35 | 31 | 30
Participants | 26 | 25 | 38 | 30 | 25 | 26 | 23

14. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory abnormalities included: Hematology (Hemoglobin [hgb], hematocrit, erythrocytes [ery]: <0.8*lower limit of normal [LLN]; reticulocytes, reticulocytes/ery: <0.5*LLN, >1.5*upper LN [ULN]; ery mean corpuscular volume [EMC], EMC hgb: <0.9*LLN, >1.1*ULN; platelet: >1.75 ULN; lymphocytes, neutrophils, basophils, eosinophils: <0.8* LLN, >1.2*ULN; monocytes: >1.2*ULN; activated partial thromboplastin time, prothrombin time: >1.1*ULN); Clinical chemistry (Total/direct bilirubin, glucose:>1.5*ULN; aspartate aminotransferase [AT], alanine AT, gamma glutamyl transferase: >3.0*ULN; HDL cholesterol: <0.8*LLN; urea nitrogen, creatinine, triglyceride, cholesterol, hgb A1C: >1.3*ULN; urate: >1.2*ULN; potassium: <0.9*LLN, >1.1*ULN; sodium: <0.95*LLN; calcium, bicarbonate: <0.9*LLN; creatine kinase: >2.0*ULN); Urinalysis (glucose, protein, hgb, ketones, nitrite, leukocyte esterase, urobilinogen, bilirubin: >=1; ery, leukocytes: >=20; granular, hyaline casts: >1).
Time Frame: as for outcome 13
Population: Safety population included all participants who took at least 1 dose of investigational product. Here, ''Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID
Number analyzed (Participants) | 34 | 34 | 48 | 42 | 35 | 31 | 30
Participants | 31 | 32 | 46 | 39 | 34 | 27 | 30

15. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Number of participants with clinically significant vital signs were reported in this outcome measure. Vital signs included blood pressure, and heart rate. Clinical significance in vital signs abnormalities was judged by investigator.
Time Frame: From first dose of study drug (Day 1) upto Week 48 (maximum up to approximately 50 weeks)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID
Number analyzed (Participants) | 34 | 34 | 48 | 42 | 35 | 31 | 30
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiograms (ECG) Parameters
Description: Number of participants with clinically significant ECG abnormalities were reported in this outcome measure. ECG parameters included heart rate, PR interval, QRS interval and QTcF interval.
Time Frame: From first dose of study drug (Day 1) upto Week 48 (maximum up to approximately 50 weeks)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID
Number analyzed (Participants) | 34 | 32 | 47 | 39 | 35 | 28 | 28
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) up to 4 weeks after last dose of study drug (maximum up to approximately 52 weeks)
Description: Same event may appear as both non-SAE and SAE but what is presented are distinct events. Event may be categorized as serious in 1 participant and non-serious in other, or participant may have experienced both serious and non-serious event. Safety population included all participants who took at least 1 dose of investigational product.
Arm/Group | Placebo | DGAT2i/PF-06865571 25 mg BID | DGAT2i/PF-06865571 75 mg BID | DGAT2i/PF-06865571 150 mg BID | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID | DGAT2i/PF-06865571 300 mg BID | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35 | 0/48 | 0/42 | 0/35 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/34 | 1/35 | 5/48 | 1/42 | 5/35 | 4/31 | 2/30
Other Adverse Events (participants affected / at risk) | 21/34 | 21/35 | 28/48 | 22/42 | 19/35 | 19/31 | 15/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | DGAT2i/PF-06865571 25 mg BID (N=35) | DGAT2i/PF-06865571 75 mg BID (N=48) | DGAT2i/PF-06865571 150 mg BID (N=42) | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID (N=35) | DGAT2i/PF-06865571 300 mg BID (N=31) | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID (N=30)
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Subcapsular hepatic hematoma (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | DGAT2i/PF-06865571 25 mg BID (N=35) | DGAT2i/PF-06865571 75 mg BID (N=48) | DGAT2i/PF-06865571 150 mg BID (N=42) | DGAT2i/PF-06865571 150 mg BID + ACCi/PF-05221304 5 mg BID (N=35) | DGAT2i/PF-06865571 300 mg BID (N=31) | DGAT2i/PF-06865571 300 mg BID + ACCi/PF-05221304 10 mg BID (N=30)
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 3 | 2 | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0 | 3 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 3 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 5 | 3 | 3 | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 5 | 1 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 2 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 4 | 1 | 0 | 3 | 1
Puncture site pain (General disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 1 | 3 | 1 | 1 | 1 | 1
COVID-19 (Infections and infestations) | 2 | 2 | 4 | 3 | 1 | 3 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 4 | 2 | 2 | 3 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 1 | 4 | 3 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 0 | 4 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 3 | 2 | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 4
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 1 | 2 | 2 | 3 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 | 6 | 5 | 3 | 2 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 2 | 3 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2 | 1 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3 | 3 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 2 | 0
Headache (Nervous system disorders) | 4 | 2 | 5 | 1 | 4 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 1 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT04321031/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT04321031/SAP_001.pdf